CLINICAL TRIAL: NCT06778967
Title: A Multicenter, Randomized, Active-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of GZR18 Injection in Chinese Subjects With Type 2 Diabetes Mellitus and Poor Blood Glucose Control by Metformin Monotherapy or in Combination With Sodium-dependent Glucose Transporter 2 (SGLT2) Inhibitors or Sulfonylureas
Brief Title: A Phase III Clinical Study to Evaluate the Efficacy and Safety of GZR18 Injection in Adult Type 2 Diabetes Mellitus
Acronym: Optimum 2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZR18-T2DM-302
Record Dates: First submitted 2025-01-03; First posted 2025-01-16 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GZR18 Dose 1 (Experimental): Participants will receive GZR18 subcutaneously (SC).
  Interventions: Drug: GZR18
- GZR18 Dose 2 (Experimental): Participants will receive GZR18 subcutaneously (SC).
  Interventions: Drug: GZR18
- semaglutide (Active Comparator): Participants will receive semaglutide subcutaneously (SC).
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: GZR18 — Administered SC
  Arms: GZR18 Dose 1; GZR18 Dose 2
Drug: semaglutide — Administered SC
  Arms: semaglutide

SUMMARY:
The main purpose of this study is to investigate the Efficacy and Safety of GZR18 Injection in Chinese Subjects with Type 2 Diabetes Mellitus and Poor Blood Glucose Control by Metformin Monotherapy or in Combination with Sodium-dependent Glucose Transporter 2 (SGLT2) Inhibitors or Sulfonylureas

ELIGIBILITY:
Inclusion Criteria:

* T2DM is diagnosed for at least 12 weeks according to the diagnostic criteria of diabetes mellitus issued by the World Health Organization (WHO) in 1999 and the supplementary diagnostic criteria of WHO in 2011 (HbA1c diagnosis is recommended).
* Antidiabetic drugs that meet any of the following within 8 weeks before screening:

  * A stable dose of metformin hydrochloride monotherapy at a dose of ≥ 1500 mg/day or the maximum tolerated dose ;

    * A stable dose of metformin (≥ 1500 mg/day or the maximum tolerated dose ) in combination with SGLT2 inhibitors;

      * A stable dose of metformin (≥1500 mg/day or a maximum tolerated dose < 1500 but ≥ 1000 mg/day) in combination with a stable daily dose of sulfonylureas.
* HbA1c ≥ 7.5% and ≤ 11% at screening (central laboratory).
* BG < 15 mmol/L at screening (central laboratory).

Exclusion Criteria:

* Type 1 diabetes mellitus or special type of diabetes mellitus.
* Diabetic ketoacidosis, diabetic lactic acidosis or hyperosmolar state within 6 months before screening, or diabetic ketosis at screening/before randomization.
* Severe chronic complications of diabetes (such as proliferative retinopathy or maculopathy, diabetic painful neuropathy, intermittent claudication, or diabetic foot) at screening or before randomization.
* History of acute or chronic pancreatitis and pancreatic injury before screening.
* History or relevant family history of medullary thyroid cancer, multiple endocrine neoplasia (MEN) 2A or 2B before screening.
* Any laboratory test indicator meeting the following criteria at screening or before randomization:
* Calcitonin level ≥ 50 ng/L (pg/mL) at screening.
* ALT ≥ 3.0 × upper limit of normal (ULN) or AST ≥ 3.0 × ULN or total bilirubin ≥ 2.0 × ULN.
* Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2, calculated using CKD-EPI equation (see Appendix 3).
* Fasting triglyceride (TG) ≥ 5.7 mmol/L or 500 mg/dL.
* Blood amylase or lipase > 1.5 × ULN.
* Hemoglobin ≤ 100 g/L for women and ≤ 110 g/L for men.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c)(%) | Baseline, Week 44

SECONDARY OUTCOMES:
Change from baseline in mean 7-point self-measured blood glucose (SMBG) | week 44
Proportion of subjects with salvage therapy. | week 44
Change from baseline in weight (kg) | week 44
Percent change in weight from baseline (%) | week 44
Proportion of subjects with ≥ 5% and 10% decrease in weight from baseline. | week 44
Treatment emergent adverse events (TEAEs) | week 44

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China